CLINICAL TRIAL: NCT02141165
Title: Efficacy and Cost-Effectiveness of a Super Simplified System for the Management of Patients With Sleep Apneas in Primary Healthcare.
Brief Title: Home Nasal Pressure for Sleep Apnea Management in Primary Case
Acronym: Primary
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, Juan F. Masa, MD, Sociedad Española de Neumología y Cirugía Torácica
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PI13/0238
Record Dates: First submitted 2014-02-17; First posted 2014-05-19 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
Keywords: sleep apnea; portable monitor; primary care; cost-effectiveness; OSAS
MeSH Terms: conditions — Sleep Apnea, Obstructive; Sleep Apnea Syndromes | interventions — Diagnosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Primary. (Experimental): Diagnosis, autoCPAP, follow up.
  Interventions: Device: Diagnosis, autoCPAP, follow up.
- Hospital (Active Comparator): Diagnosis, autoCPAP, follow up
  Interventions: Device: Diagnosis, autoCPAP, follow up.

INTERVENTIONS:
Device: Diagnosis, autoCPAP, follow up. — comparison between the efficacy of two protocol

SUMMARY:
Primary objectives: To determine the efficacy and cost-effectiveness of a management program for patients with obstructive sleep apnea syndrome (OSAS) carried out in primary or specialist healthcare. In the primary arm, the diagnosis and therapeutic decision will be made by means of a domiciliary nasal pressure (DNP) channel and oximetry while the specialist healthcare arm will use polysomnography (PSG) in a hospital. Patients with an intermediate-high suspicion of OSAS will be included, taking as primary variables the Epworth scale, for efficacy, and the Epworth scale and EuroQol 5D, for cost-effectiveness.

Secondary objectives: efficacy of the two SAHS management programs according to the following secondary variables: a) quality-of-life tests: FOSQ questionnaire, SF36 and analogical wellbeing scale, b) adherence to and compliance with the treatment.

DETAILED DESCRIPTION:
Design: prospective, randomized, controlled, open, parallel, non-inferiority. A total of 280 patients will be randomized for management on the basis of DNP (primary) or PSG (specialist), thereby giving rise to 4 groups: two treated and two not treated with CPAP. The former will undergo a home auto-titration. The follow-up will last 6 months and include 4 evaluations.

ELIGIBILITY:
Inclusion Criteria:

1. Snoring or apneas objectively observed during sleep by a partner;
2. Symptoms that are potentially secondary to apneas/hypopneas with an intermediate-high probability of being treated with CPAP. In operative terms, Epworth scale ≥12 or previous cardiovascular disease;
3. Age between 18 and 70 years;
4. Absence of any clinical suspicion of any other sleep pathology susceptible to coinciding with daytime sleepiness.

Exclusion Criteria:

1. Psycho-physical incapacity to complete questionnaires;
2. Documented structural or coronary heart disease uncontrolled by any medical treatment;
3. Cheyne-Stokes syndrome;
4. Patients subjected to uvulopalatopharyngoplasty;
5. Significant nasal obstruction impeding the use of CPAP;
6. Pregnancy;
7. Lack of informed consent.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 280 (Actual)
Dates: Start 2014-03 (Actual); Primary Completion 2016-04 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Efficacy of the extra- and intra-hospital programs using DNP or PSG, taking as primary variable the Epworth scale. | Before and after 6 months of follow-up

SECONDARY OUTCOMES:
Cost-effectiveness of the exta- and intra-hospital management programs using DNP or PSG, evaluated by means of the Epworth scale and EuroQol 5D. | Before and after 6 months of follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Juan F. Masa, MD, Principal Investigator — Hospital San Pedro de Alcántara. Cáceres. Spain
Locations (1):
- Juan Fernando Masa Jiménez, Cáceres, Cáceres, Spain

REFERENCES:
- [Derived] Sanchez-Quiroga MA, Corral J, Gomez-de-Terreros FJ, Carmona-Bernal C, Asensio-Cruz MI, Cabello M, Martinez-Martinez MA, Egea CJ, Ordax E, Barbe F, Barca J, Masa JF; Spanish Sleep Network and Primary Care Group. Primary Care Physicians Can Comprehensively Manage Patients with Sleep Apnea. A Noninferiority Randomized Controlled Trial. Am J Respir Crit Care Med. 2018 Sep 1;198(5):648-656. doi: 10.1164/rccm.201710-2061OC. PMID 29664672